CLINICAL TRIAL: NCT06922643
Title: Study of the Efficacy and Safety of Pegnano Plus Barivir (Ribavirin) in Treatment-naïve Patients With Chronic Hepatitis C at KienGiang General Hospital
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NNG00
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pegnano (Peginterferon alfa-2a) (Experimental)
  Interventions: Drug: Peginterferon Alfa-2A; Drug: Ribavirin Oral Product

INTERVENTIONS:
Drug: Peginterferon Alfa-2A — 180 mcg, subcutaneous injection, once weekly
  Other Names: Pegnano (Peginterferon alfa-2a)
Drug: Ribavirin Oral Product — 15 mg/kg daily, oral (1200 mg/day for body weight >80 kg)
  Other Names: Barivir

SUMMARY:
This study presents a clinical study on the efficacy and safety of Pegnano combined with Barivir (Ribavirin) in treating treatment-naïve patients with Chronic Hepatitis C at Kien Giang General Hospital. The study aims to provide affordable treatment options while evaluating the virological response and side effects associated with the therapy

DETAILED DESCRIPTION:
This study evaluates the efficacy and safety of Pegnano (Peginterferon alfa-2a) combined with Barivir (Ribavirin) in treatment-naïve patients with chronic hepatitis C (HCV). Conducted at Kien Giang General Hospital from March 2011 to March 2013, this uncontrolled clinical trial enrolled 100 outpatients aged 18-65 with HCV RNA >80 IU/mL and compensated liver disease. Patients received Pegnano (180 mcg, subcutaneous, weekly) and Barivir (15 mg/kg daily, oral) for 24 weeks (genotypes 2, 3) or 48 weeks (genotypes 1, 4, 5, 6), with possible extension to 72 weeks for genotype 1 with late virological response. The primary goal is to assess virological responses (rapid, early, end-of-treatment, and sustained at 24 weeks) by genotype and IL28B rs12979860 polymorphism, alongside safety through adverse event monitoring. Efficacy is measured via HCV RNA levels using real-time PCR, while safety is evaluated through clinical and paraclinical assessments every 4 weeks. The study aims to provide evidence for affordable HCV treatment options in Vietnam using locally produced drugs

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C.
* Age 18-65 years.
* No previous treatment with interferon or peginterferon.
* HCV RNA serum baseline >80 IU/mL.
* Compensated liver disease (total bilirubin <25.6 µmol/L, INR <1.5, serum albumin >3.4 g/dL, no ascites or hepatic encephalopathy).
* Normal hematological and biochemical parameters (hemoglobin >12 g/dL for males, >11 g/dL for females; neutrophils >1500 cells/µL; platelets >75,000 cells/µL; serum creatinine <1.5 mg/dL or <132 µmol/L).

Exclusion Criteria:

* Depression.
* Autoimmune hepatitis or other autoimmune diseases.
* Unstable hyperthyroidism or hypothyroidism.
* Severe medical conditions (e.g., hypertension, congestive heart failure, angina, uncontrolled diabetes, COPD).
* Decompensated cirrhosis.
* Co-infection with HIV or hepatitis B.
* Pregnant women or those unwilling to use effective contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2013-01-21 (Actual); Study Completion 2013-03-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegnano (Peginterferon Alfa-2a)
Started | 100
Completed | 97
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pegnano (Peginterferon Alfa-2a)
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight (kg) [Mean (Standard Deviation); unit: kg] | 62.4 (10)

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response (SVR)
Description: Percentage of patients with undetectable HCV RNA 24 weeks after treatment completion, measured by real-time reverse transcriptase PCR. In this study, the term "undetectable HCV RNA" refers to the absence of detectable Hepatitis C viral RNA in the patient's serum as measured by Real-Time reverse transcriptase PCR. This method exhibits high sensitivity and specificity, enabling the accurate quantification of HCV RNA. An 'undetectable' result indicates that the viral load was below the lower limit of detection of the assay used (negative). Virological responses were assessed at multiple time points, including week 4 (RVR), week 12 (cEVR), at the end of treatment (EOT), and 12 or 24 weeks post-treatment (SVR12, SVR24). Achieving 'undetectable HCV RNA' at these points was used to determine the effectiveness of the therapy.
  In this study, SVR and SVR24 are interchangeable.
Time Frame: 24 weeks post-treatment
Population: Total number of participants by viral genotype: 100
  * Genotype 1: 24 participants
  * Genotype 2: 13 participants
  * Genotype 6: 63 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Pegnano (Peginterferon Alfa-2a)
Number analyzed (Participants) | 100
Participants
  G1: number analyzed (Participants) | 24
  G1 | 17
  G2: number analyzed (Participants) | 13
  G2 | 10
  G6: number analyzed (Participants) | 63
  G6 | 56
  Total | 83
Statistical Analysis 1: Comparison: Pegnano (Peginterferon Alfa-2a); Test type: Other; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 6.73, 95% CI 2-sided [1.63 to 27.8]

2. Secondary Outcome: Rapid Virological Response (RVR)
Description: Percentage of patients with undetectable HCV RNA at week 4, measured by real-time reverse transcriptase PCR.
  In this study, the term "undetectable HCV RNA" refers to the absence of detectable Hepatitis C viral RNA in the patient's serum as measured by Real-Time reverse transcriptase PCR. This method exhibits high sensitivity and specificity, enabling the accurate quantification of HCV RNA. An 'undetectable' result indicates that the viral load was below the lower limit of detection of the assay used (negative). Virological responses were assessed at multiple time points, including week 4 (RVR), week 12 (cEVR), at the end of treatment (EOT), and 12 or 24 weeks post-treatment (SVR12, SVR24). Achieving 'undetectable HCV RNA' at these points was used to determine the effectiveness of the therapy.
Time Frame: Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pegnano (Peginterferon Alfa-2a)
Number analyzed (Participants) | 100
Participants
  G1: number analyzed (Participants) | 24
  G1 | 19
  G2: number analyzed (Participants) | 13
  G2 | 12
  G6: number analyzed (Participants) | 63
  G6 | 57

3. Secondary Outcome: Complete Early Virological Response (cEVR)
Description: Percentage of patients with undetectable HCV RNA at week 12 (in non-RVR patients), measured by real-time reverse transcriptas PCR.
  In this study, the term "undetectable HCV RNA" refers to the absence of detectable Hepatitis C viral RNA in the patient's serum as measured by Real-Time reverse transcriptase PCR. This method exhibits high sensitivity and specificity, enabling the accurate quantification of HCV RNA. An 'undetectable' result indicates that the viral load was below the lower limit of detection of the assay used (negative). Virological responses were assessed at multiple time points, including week 4 (RVR), week 12 (cEVR), at the end of treatment (EOT), and 12 or 24 weeks post-treatment (SVR12, SVR24). Achieving 'undetectable HCV RNA' at these points was used to determine the effectiveness of the therapy.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pegnano (Peginterferon Alfa-2a)
Number analyzed (Participants) | 100
Participants
  G1: number analyzed (Participants) | 24
  G1 | 24
  G2: number analyzed (Participants) | 13
  G2 | 13
  G6: number analyzed (Participants) | 63
  G6 | 63

4. Secondary Outcome: End of Treatment Response (ETR)
Description: Percentage of patients with undetectable HCV RNA at the end of treatment, measured by real-time PCR.
Time Frame: End of treatment: 24 weeks for genotypes 2 and 3; 48 weeks for genotypes 1, 4, 5, and 6. For genotypes 1 and 4, extend to 72 weeks if only LVR is achieved. For genotypes 2 and 3, extend to 48 weeks if non-RVR but EVR is present.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pegnano (Peginterferon Alfa-2a)
Number analyzed (Participants) | 100
Participants
  G1: number analyzed (Participants) | 24
  G1 | 22
  G2: number analyzed (Participants) | 13
  G2 | 13
  G6: number analyzed (Participants) | 63
  G6 | 62

5. Secondary Outcome: Safety (Adverse Events)
Description: Incidence and severity of clinical and paraclinical adverse events (e.g., anemia, neutropenia, depression), assessed every 4 weeks
Time Frame: Throughout treatment (up to 72 weeks) and 24 weeks post-treatment (up to week 96)
Measure: Count of Participants; unit: Participants
Arm/Group | Pegnano (Peginterferon Alfa-2a)
Number analyzed (Participants) | 100
Participants | 100

ADVERSE EVENTS:
Time Frame: Throughout treatment (up to 72 weeks) and 24 weeks post-treatment (up to week 96)
Arm/Group | Pegnano (Peginterferon Alfa-2a)
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 100/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegnano (Peginterferon Alfa-2a) (N=100)
Alopecia (Skin and subcutaneous tissue disorders) | 78
Anorexia (Metabolism and nutrition disorders) | 58
Sluggish (Gastrointestinal disorders) | 41
Insomnia (Psychiatric disorders) | 35
Chill (General disorders) | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 29
Mild pyrexia (without use of Paracetamol) (General disorders) | 22
Moderate Pyrexia (with use of Paracetamol) (General disorders) | 19
Fatigue (General disorders) | 22
Mild depression (Psychiatric disorders) | 13
Moderate depression (Psychiatric disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 20
Erythema at injection site (General disorders) | 11
Headache (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Hyperthyroidism with paraclinical evidences (Endocrine disorders) | 4
Hypothyroidism with paraclinical evidences (Endocrine disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No